CLINICAL TRIAL: NCT02724267
Title: A Randomized Controlled Prospective Study of Targeted Internal Radiation Therapy in Patients With Advanced Hepatocellular Carcinoma.
Brief Title: Targeted Internal Radiation Therapy in Advanced HCC Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospital, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZD201208002-P1
Record Dates: First submitted 2016-03-28; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Internal Radiation; Advanced Hepatocellular Carcinoma
Keywords: 131I-chTNT-1/B treatment
MeSH Terms: interventions — 131I-chimeric TNT-1-B monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- transcatheter arterial chemoembolization (Active Comparator): Patients will be treated with TACE only.
  Interventions: Biological: 131I-chTNT-1/B
- internal radiation group (Experimental): Patients will be treated with TACE combined with internal radiation.
  Interventions: Biological: 131I-chTNT-1/B

INTERVENTIONS:
Biological: 131I-chTNT-1/B — 29.6 MBq/kg,intravenous administration in 1 hour，1-3 course of treatment

SUMMARY:
The aim of this study is to evaluate the 131I-chTNT-1/B treatment effect and safety of individual therapy using randomized controlled study, in order to acquire the evidence of evidence-based medicine and create a new program of targeted internal radiation therapy in advanced HCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Via clinical diagnosis and confirm it is advanced hepatocellular carcinoma
2. mRECIST estimation: necrosis region in HCC
3. Negative iodine allergy test
4. Liver function ：Child-Pugh A/B

Exclusion Criteria:

1. reject to attend；
2. impossible to come to our hospital for physical examination regularly.
3. Blood clotting function hindrance; 4, Patients with apparent cardiac, pulmonary, cerebral and renal dysfunction,which may affect the treatment of liver cancer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 3 years

SECONDARY OUTCOMES:
Time to Progression | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China